CLINICAL TRIAL: NCT00764127
Title: The Development of an Eating Laboratory for Overweight Adolescents
Status: Completed | Type: Observational
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: #5217 DK074503-01; R21DK074503 (NIH)
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Adolescent Obesity
Keywords: adolescent; obesity; bariatric surgery; eating
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 10 cc (2 teaspoons) of blood will be drawn during the screening assessment to screen for medical illness.
  60 cc (12 teaspoons) of blood will be drawn from an indwelling IV catheter during the single-item meal to assay for meal-related hormones (ghrelin, leptin,cholecystokinin, insulin, peptideY). Bariatric surgery participants may have an additional 20 cc of blood taken to measure glucose responses to the meal.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Obese Control
- Normal Control
- OVERWEIGHT ADOLESCENT PATIENTS UNDERGOING BARIATRIC SURGERY

SUMMARY:
The purpose of the study is to develop methods to evaluate the eating behavior of adolescents, including overweight, normal weight, and candidates for adolescent bariatric surgery.

DETAILED DESCRIPTION:
The purpose of this study is to examine the eating behavior, meal-related perceptions and meal-related hormones in overweight adolescents, normal weight adolescents and overweight adolescents who are undergoing bariatric surgery. Subjects will be asked to consume a single-item breakfast meal of a fixed amount (Ensure) and a multiple-item meal from a luncheon buffet. During the single-item meal, subjects will fill out questionnaires assessing subjective responses to the meal (e.g. hunger, fullness, pleasantness) and blood samples will be taken before, during, and after the meal to assess hormonal responses to the meal. The multiple-item meal will permit an assessment of total caloric consumption, food and macronutrient choice and rate of eating. Overweight adolescents undergoing bariatric surgery will be asked to do the meal studies 1 to 3 months before and 3 to 6 months after their surgery. Some bariatric surgery patients will only be studied after their after their surgery.

The data gathered from these pilot subjects will be used to further develop and refine our future studies on assessing eating behavior in overweight adolescents.

ELIGIBILITY:
Inclusion Criteria:

* BMI Index Enrollment in bariatric surgery program Ages 12-18

Exclusion Criteria:

* Pervasive developmental or psychological disorder Current use of weight loss medication Clinically significant medical condition Pregnancy Food allergy to single-item meal

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2008-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Caloric intake | post-meal

CONTACTS AND LOCATIONS:
Overall Officials: Michael Devlin, M.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Derived] Sysko R, Devlin MJ, Schebendach J, Tanofsky-Kraff M, Zimmerli E, Korner J, Yanovski JA, Zitsman JL, Walsh BT. Hormonal responses and test meal intake among obese teenagers before and after laparoscopic adjustable gastric banding. Am J Clin Nutr. 2013 Nov;98(5):1151-61. doi: 10.3945/ajcn.113.061762. Epub 2013 Aug 28. PMID 23985807